CLINICAL TRIAL: NCT01485211
Title: Corneal Thickness Changes During Corneal Collagen Cross-linking With Ultraviolet-A Irradiation and Hypo-osmolar Riboflavin Solution in Thin Corneas
Brief Title: Corneal Thickness Changes During Corneal Collagen Cross-linking With Ultraviolet-A Irradiation and Riboflavin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Olhos de Goiania (Other)
Responsible Party: Principal Investigator, Joao Nassaralla, Clinical Professor, Instituto de Olhos de Goiania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BQ - 5 - 11 -ARVO
Record Dates: First submitted 2011-11-23; First posted 2011-12-05 (Estimated); Last update posted 2011-12-05 (Estimated); Status verified 2011-11

CONDITIONS: Progressive Keratoconus; Thin Corneas
Keywords: progressive keratoconus; thin corneas; cross-linking; hypo-osmolar riboflavin
MeSH Terms: interventions — Riboflavin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- crosslinking with hypoosmolar riboflavin (Experimental): Riboflavin and UVA-induced corneal cross-linking increases the stability of keratoconic corneas. The current inclusion criteria require a minimum stromal thickness of 400 µm. Hypo-osmolar riboflavin solution increases the stromal thickness before CXL in cases with preoperatively thin corneas.
  Interventions: Drug: cross-linking with hypo-osmolar riboflavin

INTERVENTIONS:
Drug: cross-linking with hypo-osmolar riboflavin — Hipo-osmolar riboflavin was applied every 20 seconds until the TCT reached 400µm. UVA irradiation was performed for 30 min. Pachymetry was recorded at the thinnest point of the cornea preoperatively, after epithelial removal, after iso-osmolar riboflavin, after hypo-osmolar riboflavin, after UVA irradiation, and at 1, 6 and 12 months.
  Other Names: Riboflavin; UVA radiation

SUMMARY:
The purpose of this study is to evaluate the corneal pachymetric variations during and after corneal collagen cross-linking (CXL) treatment with ultraviolet-A irradiation (UVA) and hypo-osmolar riboflavin solution in thin corneas.

DETAILED DESCRIPTION:
To evaluate the corneal pachymetric variations during and after corneal collagen cross-linking (CXL) treatment with ultraviolet-A irradiation (UVA) and hypo-osmolar riboflavin solution in thin corneas.

Eighteen eyes of 18 patients, 11 men and 7 women, with progressive keratoconus and thinnest corneal thickness (TCT) less than 400µm were included in this study.

After the epithelium removal, iso-osmolar riboflavin was applied to the cornea every 3 minutes (30 min). Hipo-osmolar riboflavin was then applied every 20 seconds until the TCT reached 400µm. UVA irradiation was performed for 30 min. Pachymetry was recorded at the thinnest point of the cornea preoperatively, after epithelial removal, after iso-osmolar riboflavin, after hypo-osmolar riboflavin, after UVA irradiation, and at 1, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Progressive Keratoconus
* thin corneas

Exclusion Criteria:

* Contact lens use for less than 3 weeks
* Non progressive keratoconus
* Thinest corneal thickness above 400 micra

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Corneal thickness changes during corneal collagen cross-linking with ultraviolet-A irradiation and hypo-osmolar riboflavin solution in thin corneas | Pachymetry was recorded at the thinnest point of the cornea preoperatively, after epithelial removal, after iso-osmolar riboflavin, after hypo-osmolar riboflavin, after UVA irradiation, and at 1, 6 and 12 months.
  To evaluate the corneal pachymetric variations during and after corneal collagen cross-linking treatment with ultraviolet-A irradiation and hypo-osmolar riboflavin solution in thin corneas with progressive keratoconus.

CONTACTS AND LOCATIONS:
Overall Officials: Belquiz A Nassaralla, MD, PhD, Study Chair — Instituto de Olhos de Goiania

REFERENCES:
- [Derived] Nassaralla BA, Vieira DM, Machado ML, Figueiredo MN, Nassaralla JJ Jr. Corneal thickness changes during corneal collagen cross-linking with UV-A irradiation and hypo-osmolar riboflavin in thin corneas. Arq Bras Oftalmol. 2013 May-Jun;76(3):155-8. doi: 10.1590/s0004-27492013000300005. PMID 23929075